CLINICAL TRIAL: NCT02279264
Title: Product Validation Study of RightSpot Infant pH Indicator for Rapid Bedside Verification of Proper Nasogastric (NG) Tube Placement in Newborn Intensive Care (NICU) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RightBio Metrics (Industry)
Responsible Party: Sponsor
Other Study IDs: RBM-2014-001
Record Dates: First submitted 2014-09-26; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Establish Normative pH Values in Neonates
Keywords: ph; RightSpot Infant; Feeding Tube; RightBio Metrics; placement; Nasogastric Tube; NG; infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: RightSpot Infant pH Indicator — pH indicator
  Other Names: RightBio Metrics; RSI001

SUMMARY:
Objectives:

1. To validate the accuracy of pH measurements of gastric fluid by comparing the readings from the RightSpot Infant pH Indicator to a standard clinically approved pH monitor
2. To determine what percentage of time the RightSpot Infant pH Indicator could have been used to determine the proper placement of the NG tube prior to feedings
3. To establish normative pH values for neonates

DETAILED DESCRIPTION:
RightBio Metrics has developed an indicator that rapidly checks gastric pH by aspirating gastric contents into the indicator through a nasogastric (NG) or orogastric (OG), causing a color change on the indicator. The color change represents various pH levels. Most Newborn Intensive Care Units require that NG/OG placement be confirmed after initial insertion and prior to any use. The purpose of this study is to validate the accuracy of pH measurement of gastric fluid by comparing the reading from the RightSpot Infant pH Indicator to a standard clinically approved pH monitor, and to determine what percentage of time the RightSpot Infant pH Indicator could have been used to determine the proper placement of the NG/OG tube prior to use. The gastric pH measurements will be analyzed to determine the normative pH values for neonates.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the Newborn Intensive Care Unit with an NG Tube

Exclusion Criteria:

* Infants with congenital or genetic abnormalities
* Infants with gastroschesis
* Infants with upper airway abnormalities
* Infants receiving any supplement or medication know to alter pH gastric contents
* Infants receiving Enfamil liquid human milk fortification
* Infant who are NPO status

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants in the Newborn Intensive Care Unit with an NG Tube
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
To compare the gastric pH measurement obtained from the RightSpot Indicator to the gastric pH measurement obtained from an approved pH monitor to determine the agreement and accuracy of the two modes of measurements. | 12 weeks
To determine the percentage of samples obtained by the RightSpot pH Indicator that could have been used to assist in determining proper placement of the NG tube prior to use. (% of collected samples vs. uncollected) | 12 weeks
To determine the percentage of samples obtained by the RightSpot pH Indicator that could have been used in determining proper placement of the NG tube prior to use.(% of sample accuracy) | 12 weeks
The gastric pH measurements will be collected and analyzed to determine the normative pH values for neonates | 12 weeks

SECONDARY OUTCOMES:
Gestation age at birth | 12 weeks
Adjusted gestational age at the time of testing | 12 weeks
Infants weight at the time of testing | 12 weeks
Time infant last ate | 12 weeks
Residual amount (ml) at the time of testing | 12 weeks
pH reading from gastric secretions | 12 weeks
Medications given which effect pH of gastric contents | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Banner Good Samaritan, Phoenix, Arizona, United States